CLINICAL TRIAL: NCT02190721
Title: A Multicenter, Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, Efficacy, and Immunogenicity of Daily Subcutaneous Administration of 5 ?g/kg Tbo-filgrastim in Infants, Children and Adolescents With Solid Tumors Without Bone Marrow Involvement
Brief Title: A Study to Evaluate 5 μg/kg Tbo-filgrastim in Infants, Children and Adolescents With Solid Tumors Without Bone Marrow Involvement
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XM02-ONC-201; 2014-001772-55 (EudraCT Number)
Record Dates: First submitted 2014-07-11; First posted 2014-07-15 (Estimated); Results first posted 2018-07-31 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Neutropenia
Keywords: Neutropenia
MeSH Terms: conditions — Neutropenia | interventions — Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- tbo-filgrastim (Experimental): Patients will receive subcutaneous doses of tbo-filgrastim 5 μg/kg body weight daily; each daily dose, to be administered at the investigative site
  Interventions: Drug: tbo-filgrastim

INTERVENTIONS:
Drug: tbo-filgrastim — 5 μg/kg

SUMMARY:
The purpose of the study is to evaluate the safety, pharmacokinetics, pharmacodynamics, and efficacy of daily subcutaneous administration of 5 μg/kg tbo-filgrastim in infants, children and adolescents with solid tumors without bone marrow involvement.

ELIGIBILITY:
Inclusion:

1. Male or female infants, children and adolescents aged 1 month to <16 years.
2. Patients with solid tumors without bone marrow involvement, who are scheduled to receive myelosuppressive CTX.
3. Body weight ≥5 kg.
4. Patients must have an initial diagnosis and histologic proof of their malignancy. All enrolled subjects should have signed consent for a CTX regimen that is known to be myelotoxic, with counts expected to drop below the absolute neutrophil count (ANC) of 0.5 × 109/L for at least 3 days. These regimens would include at least one of the following:

   * Etoposide
   * doxorubicin
   * ifosfamide
   * cyclophosphamide
5. ANC and platelet count: Patients must have an ANC >1 × 109/L and a platelet count >100 × 109/L to be eligible for therapy at the start of CTX.
6. Normal cardiac, renal, and hepatic function.
7. All subjects must have a life expectancy of 12 weeks or more.
8. Performance Status: Lansky performance score >60 (age 1 to <16 years).

   * More criteria may apply, please contact the investigator for more information.

Exclusion:

1. Bone marrow involvement.
2. Active myelogenous leukemia or history of myelogenous leukemia.
3. Previous treatment with colony-stimulating factors (granulocyte colony-stimulating factor [G-CSF], granulocyte-macrophage colony-stimulating factor, interleukin 11 [IL-11]) less than 6 weeks prior to study entry.
4. History of congenital neutropenia or cyclic neutropenia.
5. Pregnant or nursing female patients.
6. Fertile patients who do not agree to use highly reliable contraceptive measures Prior bone marrow or stem cell transplant, or prior radiation to ≥25% of bone marrow within the 4 weeks prior to the first tbo-filgrastim dose.
7. Ongoing active infection or history of infectious disease within 2 weeks prior to the screening visit.
8. Treatment with lithium at screening or planned during the study

   * More criteria may apply, please contact the investigator for more information.

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2015-05-12 (Actual); Primary Completion 2017-04-04 (Actual); Study Completion 2017-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (33):
- United States (7):
  - Teva Investigational Site 12958, Long Beach, California
  - Teva Investigational Site 12951, Los Angeles, California
  - Teva Investigational Site 12954, Jackson, Mississippi
  - Teva Investigational Site 12953, Las Vegas, Nevada
  - Teva Investigational Site 12959, Valhalla, New York
  - Teva Investigational Site 12960, Columbus, Ohio
  - Teva Investigational Site 12957, Houston, Texas
- Bulgaria (2):
  - Teva Investigational Site 59104, Sofia
  - Teva Investigational Site 59105, Varna
- Croatia (3):
  - Teva Investigational Site 60015, Rijeka
  - Teva Investigational Site 60014, Zagreb
  - Teva Investigational Site 60016, Zagreb
- Hungary (3):
  - Teva Investigational Site 51186, Budapest
  - Teva Investigational Site 51185, Budapest
  - Teva Investigational Site 51184, Szeged
- Poland (5):
  - Teva Investigational Site 53249, Gdansk
  - Teva Investigational Site 53248, Lublin
  - Teva Investigational Site 53245, Warsaw
  - Teva Investigational Site 53246, Warsaw
  - Teva Investigational Site 53247, Wroclaw
- Romania (3):
  - Teva Investigational Site 52063, Bucharest
  - Teva Investigational Site 52064, Cluj-Napoca, Cluj
  - Teva Investigational Site 52065, Timișoara
- Russia (5):
  - Teva Investigational Site 50282, Chelyabinsk
  - Teva Investigational Site 50281, Krasnodar
  - Teva Investigational Site 50284, Moscow
  - Teva Investigational Site 50280, Saint Petersburg
  - Teva Investigational Site 50283, Volgograd
- Ukraine (5):
  - Teva Investigational Site 58147, Kharkiv
  - Teva Investigational Site 58145, Kyiv
  - Teva Investigational Site 58148, Lviv
  - Teva Investigational Site 58146, Vinnytsia
  - Teva Investigational Site 58149, Vinnytsia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 55 patients were screened for this study. Of the 55 patients screened, 50 patients at 33 investigational centers in Central and Eastern Europe met inclusion/exclusion criteria and were considered to be eligible for enrollment into the study.
Pre-assignment Details: Of the 5 patients who were not enrolled, 2 patients were excluded due to inclusion criteria not met (baseline AST elevation, baseline ANC count was too low), 2 patients were excluded due to exclusion criteria not met (ongoing active infection or history of infectious disease within 2 weeks prior to screening), and 1 patient withdrew consent.
Groups:
- Infants (1 Month to <2 Years); Children (2 to <12 Years); Adolescents (12 to <16 Years): Tbo-filgrastim administration was started at approximately 24 hours (±3 hours) after the end of the last chemotherapy (CTX) treatment in the first week of the CTX cycle. Daily dosing with tbo-filgrastim at a dose of 5 μg/kg/day of body weight continued until the expected neutrophil nadir was passed and the neutrophil count had recovered to 2.0 × 10^9/L but not longer than 14 consecutive days. An immunogenicity sample was collected 30 days and 3 months after the last tbo-filgrastim administration in the first cycle.
Period: Overall Study
Arm/Group | Infants (1 Month to <2 Years) | Children (2 to <12 Years) | Adolescents (12 to <16 Years)
Started | 2 | 30 | 18
Completed Treatment | 2 | 30 | 18
Completed 30 Day Follow-up | 2 | 29 | 18
Completed 90 Day Follow-up | 2 | 29 | 18
Completed | 2 | 29 | 18
Not Completed | 0 | 1 | 0
Not completed — Patient was out of the city | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- Total: Total of all reporting groups
Arm/Group | Infants (1 Month to <2 Years) | Children (2 to <12 Years) | Adolescents (12 to <16 Years) | Total
Number analyzed (Participants) | 2 | 30 | 18 | 50
Age, Continuous [Median (Full Range); unit: Years] | 1.65 [1.4 to 1.9] | 6.80 [2.4 to 11.5] | 13.80 [12.0 to 15.9] | 9.05 [1.4 to 15.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 13 | 6 | 20
  Male | 1 | 17 | 12 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 30 | 18 | 50
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 2 | 30 | 18 | 50
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Weight [Median (Full Range); unit: kg] | 9.90 [9.3 to 10.5] | 20.25 [12.0 to 51.1] | 53.90 [29.5 to 89.5] | 28.95 [9.3 to 89.5]
Height [Median (Full Range); unit: cm] | 78.00 [76.0 to 80.0] | 121.00 [89.0 to 163.0] | 161.00 [140.0 to 185.0] | 130.50 [76.0 to 185.0]
Body Mass Index [Median (Full Range); unit: kg/m^2] | 16.0 [16 to 16] | 15.2 [12 to 20] | 20.7 [15 to 28] | 16.4 [12 to 28]
Chemotherapy Administration [Count of Participants; unit: Participants] — The chemotherapy (CTX) regimens administered included at least etoposide, doxorubicin, ifosfamide, or cyclophosphamide. The severity group (mild/moderate/severe) of myelotoxicity of the CTX regimens administered was assigned by a group of clinical experts, based on the scientific literature (Moreau et al 2009) and clinical experience.
  Participants
    Mild | 0 | 6 | 8 | 14
    Moderate | 2 | 16 | 7 | 25
    Severe | 0 | 8 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: Participants With Adverse Events (AEs)
Description: An adverse event was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. A treatment-emergent AE (TEAE) is an AE occurring during the timeframe. A non-TEAE is any AE not considered a TEAE.
  Severity was rated by the investigator using the NCI Common Terminology Criteria for Adverse Events (NCI-CTCAE) scale where 3=severe but not life-threatening, 4=life-threatening and 5=death. Relation of AE to treatment was determined by the investigator (related=reasonable possibility). Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical intervention to prevent the previously listed serious outcomes.
Time Frame: Non-TEAE: signing of informed consent to Day -1 (last day of CTX in week 1). And > 30 days after last dose of tbo-filgrastim (Day 46+). TEAE timeframe: Day 1 (start of tbo-filgrastim) to <= 30 days after the last dose (up to Day 45)
Population: Safety analysis set. The safety analysis set included all enrolled patients who received at least 1 dose of tbofilgrastim.
Measure: Count of Participants; unit: Participants
Arm/Group | Infants (1 Month to <2 Years) | Children (2 to <12 Years) | Adolescents (12 to <16 Years)
Number analyzed (Participants) | 2 | 30 | 18
Participants
  Any adverse event | 2 | 28 | 16
  Any TEAE | 2 | 28 | 15
  Any non-TEAE | 2 | 15 | 9
  Any treatment-related TEAE | 0 | 4 | 5
  Any TEAE with NCI-CTCAE ToxicityGrade >=3 | 2 | 18 | 8
  Any trt-related TEAE with Toxicity Grade >=3 | 0 | 1 | 2
  Any serious TEAE | 0 | 9 | 3
  Any serious treatment-related TEAE | 0 | 1 | 1
  Any TEAE leading to discontinuation | 0 | 0 | 0
  Any treatment-related TEAE leading to discont | 0 | 0 | 0
  Any TEAE leading to death | 0 | 0 | 0
  Any treatment-related TEAE leading to death | 0 | 0 | 0

2. Primary Outcome: Participants With Potentially Clinically Significant Abnormal Serum Chemistry Results
Description: Serum chemistry tests included alkaline phosphatase, alanine aminotransferase (ALT), aspartate aminotransferase (AST), direct bilirubin, indirect bilirubin, total bilirubin, calcium, creatinine, gammaglutamyl transpeptidase (GGT), glucose, potassium, lactate dehydrogenase (LDH), phosphate, sodium and uric acid.
  Only tests with potentially clinically significant abnormal results are reported.
  ULN = upper limit of normal
Time Frame: Day 1 (start of tbo-filgrastim administration) up to Day 21
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Infants (1 Month to <2 Years) | Children (2 to <12 Years) | Adolescents (12 to <16 Years)
Number analyzed (Participants) | 2 | 30 | 18
Participants
  Participants with >=1 abnormality | 0 | 3 | 1
  ALT: >20 * ULN | 0 | 1 | 1
  AST: >20 * ULN | 0 | 1 | 0
  AST: >5 * ULN and <= 20 * ULN | 0 | 0 | 1
  GGT: >5 * ULN and <= 20 * ULN | 0 | 3 | 1

3. Primary Outcome: Participants With Potentially Clinically Significant Abnormal Hematology Results
Description: Hematology tests included Basophils ABS (x 10^9/L), Basophils (%), Eosinophils ABS (x 10^9/L), Eosinophils (%), Hematocrit (%), Hemoglobin (g/L), Lymphocytes Absolute Count (ABS) (x 10^9/L), Lymphocytes (%), Monocytes ABS (x 10^9/L), Monocytes (%), Neutrophils ABS (x 10^9/L), Neutrophils (%), Platelets (x 10^9/L), Red Blood Cell (RBC) (x 10^12/L), White Blood Cell (WBC) (x 10^9/L).
  Only tests with potentially clinically significant abnormal results are reported.
  ULN = upper limit of normal
Time Frame: Day 1 (start of tbo-filgrastim administration) up to Day 21
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Infants (1 Month to <2 Years) | Children (2 to <12 Years) | Adolescents (12 to <16 Years)
Number analyzed (Participants) | 2 | 30 | 18
Participants
  Participants with >=1 abnormality | 2 | 6 | 3
  Hemoglobin (g/L): <80 | 1 | 2 | 0
  Hemoglobin (g/L): increase of >40 *ULN or baseline | 0 | 0 | 1
  Lymphocytes ABS (x 10^9/L): >=0.2 and <0.5 | 0 | 3 | 0
  Neutrophils ABS (x 10^9/L): <0.5 | 1 | 1 | 1
  Neutrophils ABS (x 10^9/L): >=0.5 and <1.0 | 1 | 1 | 1
  Platelets (x 10^9/L): >=25 and <50 | 0 | 1 | 0
  White Blood Cell (WBC) (x 10^9/L):<1.0 | 0 | 1 | 0
  White Blood Cell (WBC) (x 10^9/L):>=1 and <2 | 1 | 3 | 1

4. Primary Outcome: Participants With Potentially Clinically Significant Abnormal Vital Signs
Description: Vital sign tests included Pulse Rate (bpm), Systolic BP (mmHg), Diastolic BP (mmHg), Respiratory Rate (bpm), and Temperature (°C).
  Only tests with potentially clinically significant abnormal results are reported.
Time Frame: Day 1 (start of tbo-filgrastim administration) up to Day 21
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Infants (1 Month to <2 Years) | Children (2 to <12 Years) | Adolescents (12 to <16 Years)
Number analyzed (Participants) | 2 | 30 | 18
Participants
  Participants with >=1 abnormality | 1 | 23 | 11
  Pulse Rate (bpm): change of >=15 bpm | 0 | 14 | 9
  Systolic BP (mmHg): change of >=20mmHg | 0 | 5 | 3
  Diastolic BP (mmHg): change of >=15 mmHg | 0 | 5 | 5
  Respiratory Rate (bpm): change of >=8 breaths/min | 0 | 5 | 0
  Temperature (°C): >=38.0 °C | 1 | 14 | 4

5. Primary Outcome: Participants With Potentially Clinically Significant Abnormal Electrocardiogram Results
Description: Triplicate 12-lead ECGs were conducted at screening, predose, 4 and 6 hours postdose on day 1 of tbo-filgrastim administration, and at the end-of-study visit. The ECGs were interpreted by both the investigator and a qualified physician at the central diagnostic center as normal, abnormal not clinically significant, or abnormal clinically significant. The following parameters were measured/derived for each ECG assessment: heart rate, PR interval, RR interval, QT interval, corrected QT interval according to Fridericia's formula (QTcF), corrected QT interval according to Bazett's formula (QTcB), QRS duration, and QRS axis.
  The count of participants with potentially clinically significant ECG findings is reported.
Time Frame: Day 1 (start of tbo-filgrastim administration) pre-dose, 4 hours post dose and 6 hours post dose; Day 21 (end of study visit)
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Infants (1 Month to <2 Years) | Children (2 to <12 Years) | Adolescents (12 to <16 Years)
Number analyzed (Participants) | 2 | 30 | 18
Participants | 0 | 0 | 0

6. Primary Outcome: Participants With Negative Shifts From Baseline to End of Study in Physical Exam Findings
Description: Physical examination was performed at screening and at the end-of-study visit. The following body systems were marked as normal or abnormal and if abnormal, whether clinically significant: Head, ears, eyes, nose and throat (HEENT), chest and lungs, heart, abdomen, skin, lymph nodes and neurological.
  Any physical examination finding that is judged by the investigator as a clinically significant change (worsening) compared with a baseline value were considered as an adverse event.
  Counts of participants with a negative shift from baseline in any of the body systems (including shifts from normal to abnormal, not clinically significant) are presented.
Time Frame: Baseline: Day -21, Day 21 (end of study visit)
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Infants (1 Month to <2 Years) | Children (2 to <12 Years) | Adolescents (12 to <16 Years)
Number analyzed (Participants) | 2 | 30 | 18
Participants
  HEENT | 0 | 0 | 0
  Chest and lungs | 0 | 0 | 0
  Heart | 0 | 0 | 0
  Abdomen | 0 | 0 | 0
  Skin | 0 | 1 | 0
  Lymph nodes | 0 | 0 | 0
  Neurological | 0 | 0 | 0

7. Primary Outcome: Participants With Injection Site Reactions to Tbo-Filgrastim Administration
Description: Using Local Tolerability Assessment Scale ranging from Pain severity 0 (Absent) to 3 (Spontaneously painful)
Time Frame: Day 1 (start of tbo-filgrastim administration) up to Day 14
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Infants (1 Month to <2 Years) | Children (2 to <12 Years) | Adolescents (12 to <16 Years)
Number analyzed (Participants) | 2 | 30 | 18
Participants
  Surface ecchymosis | 2 | 7 | 2
  Surface erythema/redness | 2 | 2 | 0
  Induration | 0 | 1 | 0
  Pain at the injection site | 0 | 0 | 0

8. Primary Outcome: Participants With Negative Shifts From Baseline to End of Study in Spleen Sonography Findings
Description: The investigator assessed spleen sonography findings as normal, abnormal not clinically significant, or abnormal clinically significant.
  Data representing counts of participants with a negative shift from baseline in spleen sonography findings (including shifts from normal to abnormal, not clinically significant) are presented.
Time Frame: Baseline: Day -21, Day 21 (end of study visit)
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Infants (1 Month to <2 Years) | Children (2 to <12 Years) | Adolescents (12 to <16 Years)
Number analyzed (Participants) | 2 | 30 | 18
Participants | 0 | 0 | 0

9. Primary Outcome: Participants Who Were Alive at the 90 Day Follow-Up
Description: Summary of participant survival at 90 day follow-up.
Time Frame: 90 days post end of study visit (111 days from start of tbo-filgrastim administration)
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Infants (1 Month to <2 Years) | Children (2 to <12 Years) | Adolescents (12 to <16 Years)
Number analyzed (Participants) | 2 | 30 | 18
Participants | 2 | 30 | 18

10. Secondary Outcome: Participants With Positive Immunogenicity Findings Tested at Four Study Timepoints
Description: Blood was drawn for the assessment of anti-drug antibody (ADA) at screening, at the end-of-study visit, and at 30 and 90 days after the last administration of tbo-filgrastim in chemotherapy (CTX) cycle 1.
  The main endpoint from the assessment was the presence of antibodies in the sample, reported as positive or negative. Participants with positive results are summarized.
Time Frame: Baseline (Day -21), Day 21 (end of study visit), Day 51 (30 Day follow-up) and Day 111 (90 Day follow-up)
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Infants (1 Month to <2 Years) | Children (2 to <12 Years) | Adolescents (12 to <16 Years)
Number analyzed (Participants) | 2 | 30 | 18
Participants
  Screening | 0 | 0 | 0
  End of Study visit | 0 | 0 | 0
  30 Day Follow-up | 0 | 0 | 0
  90 Day Follow-up | 0 | 0 | 0

11. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of Tbo-Filgrastim
Time Frame: Within 1 hour before the tbo-filgrastim dose and at 2, 4, 6, 8, and 12 hours after the tbo-filgrastim dose on Day 1
Population: Pharmacokinetic (PK) analysis set
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Infants (1 Month to <2 Years) | Children (2 to <12 Years) | Adolescents (12 to <16 Years)
Number analyzed (Participants) | 2 | 29 | 18
pg/mL | 26087.95 (8647.562) | 20048.27 (9232.446) | 19032.60 (11086.273)

12. Secondary Outcome: Time to Maximum Observed Serum Concentration (Tmax) of Tbo-Filgrastim
Time Frame: Within 1 hour before the tbo-filgrastim dose and at 2, 4, 6, 8, and 12 hours after the tbo-filgrastim dose on Day 1
Population: PK analysis set
Measure: Median (Full Range); unit: Hours
Arm/Group | Infants (1 Month to <2 Years) | Children (2 to <12 Years) | Adolescents (12 to <16 Years)
Number analyzed (Participants) | 2 | 29 | 18
Hours | 6.00 [6.0 to 6.0] | 4.07 [3.9 to 8.0] | 4.00 [3.9 to 8.0]

13. Secondary Outcome: Area Under The Serum Concentration-Time Curve From Time 0 To Time Of Last Quantifiable Concentration (AUClast)
Time Frame: Within 1 hour before the tbo-filgrastim dose and at 2, 4, 6, 8, and 12 hours after the tbo-filgrastim dose on Day 1
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: hr*pg/mL
Arm/Group | Infants (1 Month to <2 Years) | Children (2 to <12 Years) | Adolescents (12 to <16 Years)
Number analyzed (Participants) | 2 | 29 | 18
hr*pg/mL | 187889.69 (80122.148) | 142124.91 (63127.420) | 127447.08 (73894.137)

14. Secondary Outcome: Area Under The Serum Concentration-Time Curve From Time 0 To 12 Hours Postdose (AUC0-12)
Time Frame: Within 1 hour before the tbo-filgrastim dose and at 2, 4, 6, 8, and 12 hours after the tbo-filgrastim dose on Day 1
Population: PK analysis set. In 4 participants, serum concentrations of tbo-filgrastim were not obtained through 12 hours and as a result, AUC0-12 could not be calculated.
Measure: Mean (Standard Deviation); unit: hr*pg/mL
Arm/Group | Infants (1 Month to <2 Years) | Children (2 to <12 Years) | Adolescents (12 to <16 Years)
Number analyzed (Participants) | 2 | 28 | 15
hr*pg/mL | 187889.69 (80122.148) | 144109.32 (63358.011) | 140550.22 (73648.629)

15. Secondary Outcome: AUC From Time 0 to Infinity (AUC0-inf)
Time Frame: Within 1 hour before the tbo-filgrastim dose and at 2, 4, 6, 8, and 12 hours after the tbo-filgrastim dose on Day 1
Population: PK analysis set. The 12 hour sampling duration limited the ability to characterize the terminal elimination rate of tbo-filgrastim (λz ) and related parameters (t½, AUC0-∞,-∞ %AUCex, CL/F, and Vz/F) for more than half of patients enrolled, especially those with maximum serum concentrations being achieved >= 6 hours. This included both infants.
Measure: Mean (Standard Deviation); unit: hr*pg/mL
Arm/Group | Infants (1 Month to <2 Years) | Children (2 to <12 Years) | Adolescents (12 to <16 Years)
Number analyzed (Participants) | 0 | 15 | 8
hr*pg/mL |  | 161964.32 (87205.040) | 198470.33 (80773.023)

16. Secondary Outcome: Elimination Half-life (t1/2)
Time Frame: Within 1 hour before the tbo-filgrastim dose and at 2, 4, 6, 8, and 12 hours after the tbo-filgrastim dose on Day 1
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Infants (1 Month to <2 Years) | Children (2 to <12 Years) | Adolescents (12 to <16 Years)
Number analyzed (Participants) | 0 | 15 | 8
hours |  | 2.41 (0.549) | 2.52 (0.561)

17. Secondary Outcome: Apparent Clearance (CL/F)
Time Frame: Within 1 hour before the tbo-filgrastim dose and at 2, 4, 6, 8, and 12 hours after the tbo-filgrastim dose of Day 1
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: L/hour
Arm/Group | Infants (1 Month to <2 Years) | Children (2 to <12 Years) | Adolescents (12 to <16 Years)
Number analyzed (Participants) | 0 | 15 | 8
L/hour |  | 0.98 (0.719) | 1.68 (0.748)

18. Secondary Outcome: Apparent Volume of Distribution During the Terminal Phase (Vz/F)
Time Frame: Within 1 hour before the tbo-filgrastim dose and at 2, 4, 6, 8, and 12 hours after the tbo-filgrastim dose on Day 1
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Infants (1 Month to <2 Years) | Children (2 to <12 Years) | Adolescents (12 to <16 Years)
Number analyzed (Participants) | 0 | 15 | 8
liters |  | 3.21 (1.963) | 6.13 (3.094)

19. Secondary Outcome: Percentage of the AUC0-∞ That Is Due To the Extrapolation (%AUCext)
Time Frame: Within 1 hour before the tbo-filgrastim dose and at 2, 4, 6, 8, and 12 hours after the tbo-filgrastim dose on Day 1
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: percent of AUC0-∞
Arm/Group | Infants (1 Month to <2 Years) | Children (2 to <12 Years) | Adolescents (12 to <16 Years)
Number analyzed (Participants) | 0 | 15 | 8
percent of AUC0-∞ |  | 7.97 (4.179) | 8.19 (4.424)

20. Secondary Outcome: Terminal Elimination Rate (Lambda-z)
Time Frame: Within 1 hour before the tbo-filgrastim dose and at 2, 4, 6, 8, and 12 hours after the tbo-filgrastim dose on Day 1
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | Infants (1 Month to <2 Years) | Children (2 to <12 Years) | Adolescents (12 to <16 Years)
Number analyzed (Participants) | 0 | 15 | 8
1/hr |  | .30 (0.077) | .29 (0.067)

21. Secondary Outcome: Participants With Severe Neutropenia
Description: Count of participants who had an incidence of severe neutropenia, defined as any value of absolute neutrophil count (ANC) <0.5 * 10^9/L at any time.
Time Frame: ANC blood samples collected within 1 hour before the tbo-filgrastim dose on Day 1, and on Days 5, 6, 7, 10, 12, 15 and at the end of study visit (up to Day 21)
Population: The Full Analysis Set (FAS) included all patients in the ITT population who received at least 1 dose of tbo-filgrastim and had at least 1 post baseline efficacy assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Infants (1 Month to <2 Years) | Children (2 to <12 Years) | Adolescents (12 to <16 Years)
Number analyzed (Participants) | 2 | 30 | 18
Participants
  Participants with event | 1 | 19 | 6
  Participants without event | 1 | 11 | 12

22. Secondary Outcome: Duration of Severe Neutropenia
Description: The duration of severe neutropenia was derived by counting the number of days with absolute neutrophil count (ANC) values <0.5 * 10^9/L.
Time Frame: as for outcome 21
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Infants (1 Month to <2 Years) | Children (2 to <12 Years) | Adolescents (12 to <16 Years)
Number analyzed (Participants) | 2 | 30 | 18
days | 1.5 (2.12) | 2.5 (2.46) | 0.7 (1.14)

23. Secondary Outcome: Area Under The Serum Drug Concentration By Time Curve Of Absolute Neutrophil Count (AUC ANC)
Time Frame: as for outcome 21
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: *10^9/L * days
Arm/Group | Infants (1 Month to <2 Years) | Children (2 to <12 Years) | Adolescents (12 to <16 Years)
Number analyzed (Participants) | 2 | 30 | 18
*10^9/L * days | 20.465 (6.1235) | 53.931 (44.8741) | 87.098 (61.1857)

24. Secondary Outcome: Absolute Neutrophil Count (ANC) Nadir
Description: ANC nadir (measured in 10^9/L) is the lowest ANC recorded.
Time Frame: as for outcome 21
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: *10^9/L
Arm/Group | Infants (1 Month to <2 Years) | Children (2 to <12 Years) | Adolescents (12 to <16 Years)
Number analyzed (Participants) | 2 | 30 | 18
*10^9/L | 0.490 (0.4808) | 0.851 (1.3633) | 0.832 (0.6358)

25. Secondary Outcome: Time to Absolute Neutrophil Count (ANC) Nadir From Beginning of Tbo-filgrastim Administration
Time Frame: as for outcome 21
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Infants (1 Month to <2 Years) | Children (2 to <12 Years) | Adolescents (12 to <16 Years)
Number analyzed (Participants) | 2 | 30 | 18
days | 3.0 (4.24) | 6.9 (2.55) | 7.3 (2.72)

26. Secondary Outcome: Time to Absolute Neutrophil Count (ANC) Nadir From Beginning of Chemotherapy
Time Frame: as for outcome 21
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Infants (1 Month to <2 Years) | Children (2 to <12 Years) | Adolescents (12 to <16 Years)
Number analyzed (Participants) | 2 | 30 | 18
days | 6.5 (2.12) | 10.3 (2.86) | 11.2 (2.31)

27. Secondary Outcome: Time to ANC Recovery To ≥1.0 * 10^9/L From ANC Nadir
Time Frame: as for outcome 21
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Infants (1 Month to <2 Years) | Children (2 to <12 Years) | Adolescents (12 to <16 Years)
Number analyzed (Participants) | 2 | 30 | 18
days | 10.0 (7.07) | 2.2 (2.02) | 1.0 (1.19)

28. Secondary Outcome: Time to ANC Recovery To ≥2.0 * 10^9/L From ANC Nadir
Time Frame: as for outcome 21
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Infants (1 Month to <2 Years) | Children (2 to <12 Years) | Adolescents (12 to <16 Years)
Number analyzed (Participants) | 2 | 30 | 18
days | 13.0 (2.83) | 3.0 (3.09) | 2.8 (2.09)

29. Secondary Outcome: Time to ANC Recovery To ≥1.0 * 10^9/L From Start of Tbo-filgrastim Administration
Time Frame: as for outcome 21
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Infants (1 Month to <2 Years) | Children (2 to <12 Years) | Adolescents (12 to <16 Years)
Number analyzed (Participants) | 2 | 30 | 18
days | 13.0 (2.83) | 7.3 (4.43) | 5.1 (5.30)

30. Secondary Outcome: Time to ANC Recovery To ≥2.0 * 10^9/L From Start of Tbo-filgrastim Administration
Time Frame: as for outcome 21
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Infants (1 Month to <2 Years) | Children (2 to <12 Years) | Adolescents (12 to <16 Years)
Number analyzed (Participants) | 2 | 30 | 18
days | 16.0 (1.41) | 8.1 (5.20) | 10.2 (4.22)

31. Secondary Outcome: Time to ANC Recovery To ≥1.0 * 10^9/L From Start of Chemotherapy
Time Frame: as for outcome 21
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Infants (1 Month to <2 Years) | Children (2 to <12 Years) | Adolescents (12 to <16 Years)
Number analyzed (Participants) | 2 | 30 | 18
days | 16.5 (4.95) | 10.2 (5.98) | 7.4 (7.09)

32. Secondary Outcome: Time to ANC Recovery To ≥2.0 * 10^9/L From Start of Chemotherapy
Time Frame: as for outcome 21
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Infants (1 Month to <2 Years) | Children (2 to <12 Years) | Adolescents (12 to <16 Years)
Number analyzed (Participants) | 2 | 30 | 18
days | 19.5 (0.71) | 11.0 (6.52) | 14.0 (3.73)

33. Secondary Outcome: Participants With Febrile Neutropenia During the First Cycle of Chemotherapy
Description: Febrile neutropenia was defined as an axillary or external ear temperature >38.3°C (100.94°F) or 2 consecutive readings >37.8°C (100.04°F) at least 2 hours apart and an ANC <0.5 * 10^9/L. The efficacy variable was evaluated for up to 21 days from the start of the first cycle of chemotherapy.
Time Frame: (relative to tbo-filgrastim therapy) Days -7 to Day 14
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Infants (1 Month to <2 Years) | Children (2 to <12 Years) | Adolescents (12 to <16 Years)
Number analyzed (Participants) | 2 | 30 | 18
Participants
  Participants with event | 1 | 9 | 3
  Participants without event | 1 | 21 | 15

ADVERSE EVENTS:
Time Frame: Day 1 (start of tbo-filgrastim administration) to <= 30 days after the last dose (up to Day 45)
Arm/Group | Infants (1 Month to <2 Years) | Children (2 to <12 Years) | Adolescents (12 to <16 Years)
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/30 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/2 | 9/30 | 3/18
Other Adverse Events (participants affected / at risk) | 2/2 | 27/30 | 15/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infants (1 Month to <2 Years) (N=2) | Children (2 to <12 Years) (N=30) | Adolescents (12 to <16 Years) (N=18)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 4 (5) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 4 (6) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (2)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hangnail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infants (1 Month to <2 Years) (N=2) | Children (2 to <12 Years) (N=30) | Adolescents (12 to <16 Years) (N=18)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 12 (20) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 5 (5) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 6 (11) | 3 (3)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (3)
Neutropenia (Blood and lymphatic system disorders) | 2 (6) | 16 (34) | 9 (16)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (5) | 8 (16) | 4 (5)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Abdominal rigidity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (2)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 5 (6) | 3 (6)
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 3 (3) | 3 (3)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 2 (10)
Hypogammaglobulinaemia (Immune system disorders) | 0 (0) | 0 (0) | 3 (6)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (2)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (3) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 2 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (4)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Neurotoxicity (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2016-02-24): https://cdn.clinicaltrials.gov/large-docs/21/NCT02190721/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-26): https://cdn.clinicaltrials.gov/large-docs/21/NCT02190721/SAP_001.pdf